CLINICAL TRIAL: NCT06931015
Title: Staging Heart Failure With Preserved Ejection Fraction by Assessing Cardiac Chamber Involvement With Echocardiography
Brief Title: Staging Heart Failure With Preserved Ejection Fraction
Acronym: StageHFpEF
Status: Not yet recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 05-22
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Cardiovascular Diseases; Heart Failure
Keywords: HFpEF; Staging; Classification; Echocardiography
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HFpEF Stage 1: Isolated left ventricle involvement: Established if patients meet the criteria of Stage 1, according to the proposed classification, which are:
  * LVMI >115 g/m2 in men/ and >95 g/m2 in women or
  * Relative wall thickness (RWT) >0.42 or
  * Elevated LV filling pressures at rest (E/e' >9)
  doi.org/10.15420/ecr.2024.31
  Interventions: Other: No interventions
- HFpEF Stage 2: Left atrial myopathy: Stage 1 criteria, plus:
  * LAVI >34 ml/m2, if sinus rhythm or
  * AF
  Interventions: Other: No interventions
- HFpEF Stage 3: Pulmonary vasculature involvement: Stage 1-2 criteria, plus:
  * Pulmonary artery systolic pressure (PASP) >35 mmHg and/or
  * Tricuspid regurgitation (TR) velocity >2.8 m/s
  Interventions: Other: No interventions
- HFpEF Stage 4: Right chambers involvement: Stage 1-3 criteria, plus:
  * Fractional area change (FAC) <35% or
  * S' <9.5 cm/s and/or
  * Tricuspid annular plane systolic excursion (TAPSE) <17 mm and/or
  * Right atria (RA) volume index (>39 ml/m2 in men/ >33 ml/m2 for women)
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is considered a systemic condition in which the prevalence of cardiovascular, metabolic, pulmonary and renal conditions determine the extent of cardiac involvement. Numerous attempts have been made to phenotype HFpEF, but patients still lack a clinically and/or prognostically relevant approach.

Progressive cardiac deterioration in HFpEF appears to be associated with a worse prognosis. However, no attempt has been made to classify the extent of cardiac involvement in HFpEF. Investigators proposed the concept of HFpEF staging according to the extent of cardiac involvement identified by transthoracic echocardiography: Stage 1: isolated left ventricular involvement; Stage 2: left atrial myopathy; Stage 3: pulmonary vasculature involvement; and Stage 4: right chambers involvement.

The study aims to investigate the associations between the proposed stages and clinical outcomes in HFpEF patients.

DETAILED DESCRIPTION:
HFpEF is a major global public health concern due to increasing incidence and prevalence, poor prognosis and limited availability of disease-modifying therapy. The management of HFpEF and the development of novel treatments are complicated due to the heterogeneous nature of the disease, which presents multiple clinical phenotypes. Each is characterised by a unique combination of cardiac and non-cardiac comorbidities such as hypertension, obesity, type 2 diabetes, chronic kidney disease, chronic obstructive pulmonary disease and others. Numerous attempts have been made to phenotype HFpEF, but patients still lack a clinically and/or prognostically relevant approach.

Looking beyond the phenotypes, HFpEF is considered a systemic condition in which the prevalence of cardiovascular, metabolic, pulmonary and renal conditions determine the extent of cardiac involvement. Progressive cardiac deterioration in HFpEF appears to be associated with a worse prognosis. However, no attempt has been made to classify the extent of cardiac involvement in HFpEF.

Investigators proposed the concept of HFpEF staging according to the extent of cardiac involvement identified by transthoracic echocardiography (TTE), which includes four stages: Stage 1: isolated left ventricular involvement; Stage 2: left atrial myopathy; Stage 3: pulmonary vasculature involvement; and Stage 4: right chambers involvement. Emerging data suggest that every subsequent cardiac chamber deterioration could be of prognostic value.

The study aims to investigate the associations between the proposed stages and clinical outcomes in HFpEF patients.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age, male and female
2. Heart failure symptoms, New York Heart Association (NYHA) II- III
3. Left ventricular ejection fraction (LVEF) > 50% documented by echocardiography at screening
4. One of the following scenarios:

   A) At screening, N-terminal pro-B-type natriuretic peptide (NT-proBNP) ≥300 pg/mL (sinus rhythm) or ≥600 pg/mL (if AF) and echocardiographic criteria see #5

   B) Previously confirmed HFpEF in combination with a history of hospitalization for HFpEF decompensation >30 days before screening defined as the presence of dyspnea and 2 of the following:
   * Rales on chest auscultation or sings of congestion on X-ray/CT scan
   * Peripheral Oedema
   * Elevated NT-proBNP ≥300 pg/mL (sinus rhythm) or ≥600 pg/mL (if AF)
5. Structural and/or functional abnormalities of heart, at least one of the following:

   * Left atrial volume index (LAVI) >34 mL/m2 (if AF >40 mL/m2)
   * Left ventricular mass index (LVMI) =115 g/m2 for males and =95 g/m2 for females
   * Relative wall thickness > 0.42
   * E/e' ratio at rest >9
6. Stable doses of oral loop diuretics, if prescribed
7. Ability to provide informed consent

Exclusion Criteria:

* Any prior measurements of LVEF <50%
* Established diagnosis of infiltrative (amyloidosis etc.), hypertrophic cardiomyopathy, muscular dystrophies, complex congenital heart disease, active myocarditis or pericardial constriction
* Planned interventions, including major cardiac surgery, percutaneous coronary intervention (PCI), transcatheter aortic valve implantation (TAVI), or implantation of cardiac resynchronization therapy
* Elective PCI or atrial fibrillation ablation within 30 days before visit
* Moderate and severe valve stenosis and more than mild primary valve regurgitation
* Acute myocardial infarction in the last 3 months, cardiac surgery, pulmonary embolism or cerebrovascular accident within the last six months
* Candidates for heart transplantation
* Secondary hypertension
* Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease
* Any active cancer
* Infective endocarditis
* Alcoholic cirrhosis
* End-stage kidney disease
* Any other condition judged by the investigator that could account for heart failure symptoms and signs (e.g., anaemia, hypothyroidism).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HFpEF, male and female, 40 years old and over who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2028-04-13 (Estimated); Study Completion 2028-12-13 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of composite endpoint of all-cause death or HF hospitalisation | From randomisation to end of 12 months follow-up
  Measured in months

SECONDARY OUTCOMES:
Number of all-cause deaths, Cardiovascular (CV) deaths, HF hospitalisations or urgent HF visits | From randomisation to end of 12 months follow-up
  Measured as count of event
Time to occurrence of all-cause death | From randomisation to end of 12 months follow-up
  Measured in months
Time to occurrence of CV death | From randomisation to end of 12 months follow-up
  Measured in months
Time to first HF hospitalisation or urgent HF Visit | From randomisation to end of 12 months follow-up
  Measured in months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Shchendrygina, Principal Investigator — Sechenov University
Locations (1):
- A Shchendrygina, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The publication which define the concept of Staging Heart Failure with Preserved Ejection Fraction by Assessing Cardiac Chamber Involvement — https://www.ecrjournal.com/articles/staging-heart-failure-preserved-ejection-fraction-assessing-cardiac-chamber-involvement?language_content_entity=en